CLINICAL TRIAL: NCT05212675
Title: Short Daily Versus Conventional Hemodialysis for COVID-19 Patients: A Randomized Study
Brief Title: Short Daily Versus Conventional Hemodialysis for COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Assistant Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBMU-1400-10
Record Dates: First submitted 2022-01-24; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Dialysis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short daily dialysis (Other): 7 days 2hours dialysis
  Interventions: Other: Short daily dialysis
- conventional dialysis (No Intervention): 3 times weekly 4hours dialysis

INTERVENTIONS:
Other: Short daily dialysis — 7 days 2hours dialysis
  Arms: short daily dialysis

SUMMARY:
Treatment of dialysis patients involved with COVID-19 with short daily hemodialysis has been supposed to improve short term outcome. It is unclear if short daily dialysis would optimize mortality or ICU admission in routine dialysis patients with COVID-19.

Also the potential variants according with worse outcomes remain to be fully elucidated.

DETAILED DESCRIPTION:
investigators undertook a randomized trial in ESRD patients infected with COVID-19 to determine: 1) if short-daily hemodialysis is associated with a reduction in mortality and ICU admission in one weak period and; 2) the potential effective variants in worst outcome. . Paperwork for the trial was submitted to the shaheed beheshti university of medical sciences in June 2021 for registration . The protocol for this trial and supporting CONSORT checklist are available. The SBMU Ethics Board approved the study and all amendments. The study was conducted according to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients >3months on hemodialysis admitted for COVID-19

Exclusion Criteria:

* ESRD patients <3 months on hemodialysis infected with COVID-19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of randomization until the date of first documented progression or date of death
  discharged or dead
ICU add | From date of randomization until the date of first documented progression or date of death
  admission to ICU or not

CONTACTS AND LOCATIONS:
Overall Officials: Nooshin Dalili, MD, Principal Investigator — SBMU
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No